CLINICAL TRIAL: NCT00617136
Title: Perioperative Temperature Management: A Big Small Problem
Brief Title: Perioperative Temperature Management
Acronym: HOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Christa Boer, Prof.dr. C. Boer, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007/235
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Hypothermia
Keywords: Surgery; Anesthesia; Hypothermia; Temperature; Perioperative; Temperature Management
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- III (Experimental): Prewarming by HotDog
  Interventions: Device: Pre- and intraoperative warming (HotDog)
- I (Active Comparator): Intraoperative warming by Bair Hugger
  Interventions: Device: Intraoperative warming (Bair Hugger)
- II (Active Comparator): Intraoperative warming by HotDog
  Interventions: Device: Intraoperative warming (HotDog)

INTERVENTIONS:
Device: Intraoperative warming (Bair Hugger) — Intraoperative warming
  Arms: I
Device: Pre- and intraoperative warming (HotDog) — Pre- and intraoperative warming by HotDog
  Arms: III
Device: Intraoperative warming (HotDog) — Intraoperative warming
  Arms: II

SUMMARY:
The investigators aim to investigate the effects of prewarming of patients undergoing elective orthopedic surgery on intraoperative temperature control and blood loss and postoperative patient discomfort and glucose and insulin levels.

DETAILED DESCRIPTION:
Hypothermia, defined as a core temperature below 36 degrees celsius, is commonly seen in patients undergoing surgery. Intraoperative hypothermia is related to postoperative patient discomfort, impaired wound healing, increased blood loss, anxiety and disturbances in glucose and insulin levels. Prewarming of patients prior to surgery may result in maintenance of intraoperative temperature and reduce postoperative complications. We therefore aim to investigate the effects of prewarming of patients undergoing elective orthopedic surgery on intraoperative temperature control and blood loss and postoperative patient discomfort and glucose and insulin levels.

Objective of the study:

Does preoperative heating of patients undergoing elective orthopedic surgery reduce the incidence of intraoperative hypothermia and postoperative comfort and modulate postoperative glucose and insulin blood levels?

Study design:

Multi-center, prospective, randomized clinical trial.

Study population:

Patients undergoing an elective orthopedic hip- or knee replacement

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective orthopedic knee- or hip replacement
* Participation based on informed consent
* > 18 years old and < 85 years old

Exclusion Criteria:

* BMI 18.5 > x < 40
* Pregnancy
* Non elective trauma patients
* Infectious or febrile patients (> 37.5oC)
* Diabetes Mellitus
* Combined surgery
* Anemia (Hb < 4.0 mmol/l)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of perioperative hypothermia | During surgery (1 hour after start warming)

SECONDARY OUTCOMES:
Perioperative blood loss | During surgery
Patient discomfort as defined by pain, nausea and vomiting, shivering and thermal discomfort | During surgery
Postoperative glucose and insulin levels | 1 hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christa Boer, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (3):
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - Spaarne Ziekenhuis, Hoofddorp
  - Isala Klinieken, Zwolle